CLINICAL TRIAL: NCT04645030
Title: The Value of Ultralow Dosis CT and Ultrasound in the Diagnosing of Pneumonia in the Emergency Department
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: SHS-ED-11b-2020
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Respiratory Tract Infections
Keywords: Pneumonia; Ultrasound; Ultra low-dose CT
MeSH Terms: conditions — Respiratory Tract Infections; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients suspected of pneumonia: Patients suspected for pneumonia after initial evaluation by the treating physician.
  Interventions: Diagnostic Test: Ultra low-dose computer thermography; Diagnostic Test: lung ultrasound

INTERVENTIONS:
Diagnostic Test: Ultra low-dose computer thermography — The ULD-CT scan will be executed according to a standardized predeveloped technical protocol. The technical protocol will differentiate between patients with BMI <25 and >25 to insure optimal ULD-CT image quality.
Diagnostic Test: lung ultrasound — LUS will be performed by trained researchers. Before inclusion researchers preforming LUS scans, will undergo a training program and will complete 25 supervised LUS scans to be certified in LUS. At the end of the training program, researchers will be tested to insure proficiency in LUS.
  LUS will be performed according to LUS protocol with seven scanning's zones on each side; 2 anterior, 2 lateral and 3 posterior.

SUMMARY:
Pneumonia is one of the most common infections in the emergency department (ED). Nevertheless, the current diagnostic tools are often slow and inaccurate. Currently, a chest x-ray is the first choice for diagnostic imaging for pneumonia in the ED, but is inaccurate with low sensitivity and specificity, resulting in both over-and underdiagnosing of pneumonia. Alternatively, computer thermography (CT) and high-resolution CT (HR-CT) offers high diagnostic accuracy but involves significantly increased radiation to the patient, and increased costs and examination time. Lately, two alternatives to chest x-ray have emerged:

* The first is lung ultrasound (LUS) which has shown higher sensitivity and specificity for pneumonia than a chest x-ray when performed by experts. However, the diagnostic accuracy of lung ultrasound performed by novice operators in the ED still needs investigation.
* The second alternative to chest x-ray is ultra-low-dose CT (ULD-CT). A ULD-CT is a CT scan where the radiation dose is significantly reduced, while still maintaining acceptable image quality. In effect merging the high diagnostic accuracy of chest CT with the low radiation doses of chest X-ray.

The aim of this study is to investigate the diagnostic accuracy of LUS by novice operators in the ED and the diagnostic accuracy of ULD-CT thorax, in patients suspected of having pneumonia.

DETAILED DESCRIPTION:
Community-acquired pneumonia (CAP) is one of the most common infectious diseases in the emergency department (ED). In Denmark, the incidence of hospitalization is 809 per 100,000 and 30-day mortality is 13%. In 2018, 29.5 per 100.000 people died of pneumonia. An increase from 27.7 per 100,000 in 2017. CAP is usually suspected in patients with dyspnea, cough and fever, without other probable explanations or when other differential diagnosis is less likely. However often patients present with vague and uncharacteristic symptoms such as altered state of consciousness, gastrointestinal symptoms or pain. Likewise is fever not always present in the elderly. The most common CAP pathogens are Streptococcus pneumoniae, Haemophilus influenzae, and gram-negative bacilli. Other notable microbiological pathogens include viruses such as Influenza, COVID-19, parainfluenza and respiratory syncytial virus. Viruses are associated with bacterial co-infections, leading to increase mortality and complications such as admission to the ICU. Normally, when a pulmonary infection is suspected, a chest X-ray is performed. Chest x-rays have a sensitivity of 43,5% (39,4-50,8) and a specificity of 93% (92.1-93.9) for pulmonary opacities compared to CT. A chest x-ray has a sensitivity of 79% for pneumonia. Computed tomography (CT) scan of the thorax has higher diagnostic precision and results improve management but result in a correspondingly increased amount of radiation compared to chest X-ray. An ultra-low-dose CT (ULD-CT) scan of the thorax may be an alternative to CT scan. ULD-CT has a radiation dose of approx. 1.5 times greater than the radiation dose of a chest X-ray and approx. 1.5% of a CT scan. ULD-CT has shown better image quality than chest X-ray, and for acutely admitted patients with dyspnea, it has a clinical effect on both diagnosis and treatment. Like chest X-rays, basic findings on ULD-CT of the thorax can be interpreted by trained clinicians.

Ultrasound is a fast non-invasive diagnostic test, without radiation. LUS has high sensitivity and specificity, with the area under ROC (AUC) of 0.95-0.98 for pneumonia. A meta-study for the use of LUS in the diagnosis of pneumonia in the ED has shown a sensitivity of 92% (87-96%) and a specificity of 94% (87-97%). AUC was calculated at 0.97. The ultrasound operators in the meta-study were all experienced ultrasound operators. Ultrasound is an operator-dependent tool and in children, it has been demonstrated that LUS diagnostic accuracy for pneumonia, is significantly lower when performed by a novice sonographer compared to an advanced sonographer. There are few if any studies that have investigated the diagnostic accuracy of novice LUS operator, in the ED, for pneumonia.

Study goals and objectives The project is divided into two, a ULD-CT study and an LUS study. The study will aim to investigate their diagnostic capabilities in at emergency department setting.

The main objective of the ULD-CT study is to investigate and answer:

* Can ULD-CT be used to diagnose pneumonia in the emergency department?
* How is the agreement between the results from ULD-CT and results from HR-CT
* Is ULDCT more sensitive and specific than standard chest x-ray in the diagnosis of pneumonia?

The investigators hypothesize that ULD-CT can be used in the evaluation of patients with pneumonia and the sensitivity, specificity and area under the curve (AUC ) of ULD-CT is higher than a chest x-ray. The null-hypothesis is that ULD-CT is not an accurate diagnostic tool for pneumonia in the emergency department.

The main objective of the LUS study is to investigate and answer:

* Can LUS be used to diagnose pneumonia in the emergency department, with newly certified LUS operators?
* How is the agreement between the results from LUS and the results from HR-CT
* Is LUS more sensitive and specific than standard chest x-ray in the diagnosis of pneumonia?

The investigators hypothesize that LUS can be used in the evaluation of patients with pneumonia by recently certified operators and the sensitivity, specificity and AUC of LUS is higher than chest x-ray in an emergency department setting. The null-hypothesis is that LUS performed by recently certified operators is not an accurate diagnostic tool for pneumonia in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Admission to an emergency department in the study, with one of following symptoms: dyspnea, cough, expectoration.
* Indication for blood culture
* Indication for chest x-ray OR
* the treating physician suspects a pneumonia diagnosis after the first evaluation of the patient

Exclusion Criteria:

* Patients < 40 years old due to risk of cancer from the radiation
* If the attending physician considers that participation will delay a life-saving treatment or patient needs direct transfer to the intensive care unit.
* Admission within the last 14 days
* Verified COVID-19 disease within 14 days before admission
* Pregnant women
* Severe immunodeficiencies: Primary immunodeficiencies and secondary immunodeficiencies (HIV positive CD4 <200, Patients receiving immunosuppressive treatment (ATC L04A), Corticosteroid treatment (>20 mg/day prednisone or equivalent for >14 days within the last 30 days), Chemotherapy within 30 days)
* Patients < 65 who already participated once due to risk of cancer from the radiation

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults admitted to the ED will be invited to participate in the study, if the physician, receiving the patient, suspects the patient has an infection (e.g. indication for blood culture) and if the physician suspects community-acquired pneumonia. The physician will base his/her suspicion on clinical symptoms such as cough, increased sputum production, chest tightness, dyspnea and fever > 38⁰C, and indication for chest x-ray.
Sampling Method: Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic capabilities of Ultra low-dose computer thermography for pneumonia | Within 24 hours from hospital admission
  True positive, true negative, false positive and false negative for ultra low-dose computer thermography for pneumonia.
Title Diagnostic capabilities of lung ultrasound for pneumonia | Within 24 hours from hospital admission
  True positive, true negative, false positive and false negative for lunge ultrasound for pneumonia.

SECONDARY OUTCOMES:
Diagnostic capabilities of chest x-ray for pneumonia | Within 24 hours from hospital admission
  True positive, true negative, false positive and false negative for chest x-ray for pneumonia

OTHER OUTCOMES:
CURB-65 score for pneumonia severity | within 4 hours from admission
  Confusion of new onset, Blood Urea nitrogen greater than 7 mmol/L (19 mg/dL), respiratory rate of 30 breaths per minute or greater, blood pressure less than 90 mmHg systolic or diastolic blood pressure 60 mmHg or less and age 65 or older
PSI | within 4 hours from admission
  Risk classes to predict the severity of pneumonia. Scores are given based on demographics, comorbidity, clinical measurements and physical Exam Findings (<70 = Risk Class II, 71-90 = Risk Class III, 91-130 = Risk Class IV, >130 = Risk Class V)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Backer Mogensen, Principal Investigator — Institute for Regional Sundhedsforskning
Locations (1):
- Hospital of Southern Jutland, Aabenraa, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sogaard M, Nielsen RB, Schonheyder HC, Norgaard M, Thomsen RW. Nationwide trends in pneumonia hospitalization rates and mortality, Denmark 1997-2011. Respir Med. 2014 Aug;108(8):1214-22. doi: 10.1016/j.rmed.2014.05.004. Epub 2014 May 20. PMID 24898129
- [Background] Eshwara VK, Mukhopadhyay C, Rello J. Community-acquired bacterial pneumonia in adults: An update. Indian J Med Res. 2020 Apr;151(4):287-302. doi: 10.4103/ijmr.IJMR_1678_19. PMID 32461392
- [Background] MacIntyre CR, Chughtai AA, Barnes M, Ridda I, Seale H, Toms R, Heywood A. The role of pneumonia and secondary bacterial infection in fatal and serious outcomes of pandemic influenza a(H1N1)pdm09. BMC Infect Dis. 2018 Dec 7;18(1):637. doi: 10.1186/s12879-018-3548-0. PMID 30526505
- [Background] Self WH, Courtney DM, McNaughton CD, Wunderink RG, Kline JA. High discordance of chest x-ray and computed tomography for detection of pulmonary opacities in ED patients: implications for diagnosing pneumonia. Am J Emerg Med. 2013 Feb;31(2):401-5. doi: 10.1016/j.ajem.2012.08.041. Epub 2012 Oct 18. PMID 23083885
- [Background] Hagaman JT, Rouan GW, Shipley RT, Panos RJ. Admission chest radiograph lacks sensitivity in the diagnosis of community-acquired pneumonia. Am J Med Sci. 2009 Apr;337(4):236-40. doi: 10.1097/MAJ.0b013e31818ad805. PMID 19365166
- [Background] Hayden GE, Wrenn KW. Chest radiograph vs. computed tomography scan in the evaluation for pneumonia. J Emerg Med. 2009 Apr;36(3):266-70. doi: 10.1016/j.jemermed.2007.11.042. Epub 2008 Jun 20. PMID 18571356
- [Background] Claessens YE, Debray MP, Tubach F, Brun AL, Rammaert B, Hausfater P, Naccache JM, Ray P, Choquet C, Carette MF, Mayaud C, Leport C, Duval X. Early Chest Computed Tomography Scan to Assist Diagnosis and Guide Treatment Decision for Suspected Community-acquired Pneumonia. Am J Respir Crit Care Med. 2015 Oct 15;192(8):974-82. doi: 10.1164/rccm.201501-0017OC. PMID 26168322
- [Background] Brenner DJ, Hall EJ. Computed tomography--an increasing source of radiation exposure. N Engl J Med. 2007 Nov 29;357(22):2277-84. doi: 10.1056/NEJMra072149. No abstract available. PMID 18046031
- [Background] Mayo-Smith WW, Hara AK, Mahesh M, Sahani DV, Pavlicek W. How I do it: managing radiation dose in CT. Radiology. 2014 Dec;273(3):657-72. doi: 10.1148/radiol.14132328. PMID 25420167
- [Background] Kroft LJM, van der Velden L, Giron IH, Roelofs JJH, de Roos A, Geleijns J. Added Value of Ultra-low-dose Computed Tomography, Dose Equivalent to Chest X-Ray Radiography, for Diagnosing Chest Pathology. J Thorac Imaging. 2019 May;34(3):179-186. doi: 10.1097/RTI.0000000000000404. PMID 30870305
- [Background] Macri F, Greffier J, Pereira F, Rosa AC, Khasanova E, Claret PG, Larbi A, Gualdi G, Beregi JP. Value of ultra-low-dose chest CT with iterative reconstruction for selected emergency room patients with acute dyspnea. Eur J Radiol. 2016 Sep;85(9):1637-44. doi: 10.1016/j.ejrad.2016.06.024. Epub 2016 Jul 1. PMID 27501900
- [Background] Alzahrani SA, Al-Salamah MA, Al-Madani WH, Elbarbary MA. Systematic review and meta-analysis for the use of ultrasound versus radiology in diagnosing of pneumonia. Crit Ultrasound J. 2017 Dec;9(1):6. doi: 10.1186/s13089-017-0059-y. Epub 2017 Feb 27. PMID 28244009
- [Background] Long L, Zhao HT, Zhang ZY, Wang GY, Zhao HL. Lung ultrasound for the diagnosis of pneumonia in adults: A meta-analysis. Medicine (Baltimore). 2017 Jan;96(3):e5713. doi: 10.1097/MD.0000000000005713. PMID 28099332
- [Background] Orso D, Guglielmo N, Copetti R. Lung ultrasound in diagnosing pneumonia in the emergency department: a systematic review and meta-analysis. Eur J Emerg Med. 2018 Oct;25(5):312-321. doi: 10.1097/MEJ.0000000000000517. PMID 29189351
- [Background] Lichtenstein DA. Lung ultrasound in the critically ill. Ann Intensive Care. 2014 Jan 9;4(1):1. doi: 10.1186/2110-5820-4-1. PMID 24401163
- [Background] Strom JJ, Haugen PS, Hansen MP, Graumann O, Jensen MBB, Aakjaer Andersen C. Accuracy of lung ultrasonography in the hands of non-imaging specialists to diagnose and assess the severity of community-acquired pneumonia in adults: a systematic review. BMJ Open. 2020 Jun 17;10(6):e036067. doi: 10.1136/bmjopen-2019-036067. PMID 32554727
- [Background] Olgers TJ, Azizi N, Blans MJ, Bosch FH, Gans ROB, Ter Maaten JC. Point-of-care Ultrasound (PoCUS) for the internist in Acute Medicine: a uniform curriculum. Neth J Med. 2019 Jun;77(5):168-176. PMID 31264587
- [Background] Tsou PY, Chen KP, Wang YH, Fishe J, Gillon J, Lee CC, Deanehan JK, Kuo PL, Yu DTY. Diagnostic Accuracy of Lung Ultrasound Performed by Novice Versus Advanced Sonographers for Pneumonia in Children: A Systematic Review and Meta-analysis. Acad Emerg Med. 2019 Sep;26(9):1074-1088. doi: 10.1111/acem.13818. Epub 2019 Jul 16. PMID 31211896
- [Background] Lichtenstein D, Meziere G, Seitz J. The dynamic air bronchogram. A lung ultrasound sign of alveolar consolidation ruling out atelectasis. Chest. 2009 Jun;135(6):1421-1425. doi: 10.1378/chest.08-2281. Epub 2009 Feb 18. PMID 19225063
- [Background] Reissig A, Kroegel C. Sonographic diagnosis and follow-up of pneumonia: a prospective study. Respiration. 2007;74(5):537-47. doi: 10.1159/000100427. Epub 2007 Feb 27. PMID 17337882
- [Background] Huda W, Ogden KM, Khorasani MR. Converting dose-length product to effective dose at CT. Radiology. 2008 Sep;248(3):995-1003. doi: 10.1148/radiol.2483071964. PMID 18710988
- [Background] Sodickson A, Baeyens PF, Andriole KP, Prevedello LM, Nawfel RD, Hanson R, Khorasani R. Recurrent CT, cumulative radiation exposure, and associated radiation-induced cancer risks from CT of adults. Radiology. 2009 Apr;251(1):175-84. doi: 10.1148/radiol.2511081296. PMID 19332852
- [Derived] Skjot-Arkil H, Heltborg A, Lorentzen MH, Cartuliares MB, Hertz MA, Graumann O, Rosenvinge FS, Petersen ERB, Ostergaard C, Laursen CB, Skovsted TA, Posth S, Chen M, Mogensen CB. Improved diagnostics of infectious diseases in emergency departments: a protocol of a multifaceted multicentre diagnostic study. BMJ Open. 2021 Sep 30;11(9):e049606. doi: 10.1136/bmjopen-2021-049606. PMID 34593497